CLINICAL TRIAL: NCT02482194
Title: Autologous Transplantation of Bone Marrow Mesenchymal Stem Cells in Patients of Spinal Cord Injury-Phase I Clinical Trial
Brief Title: Autologous Mesenchymal Stem Cells Transplantation for Spinal Cord Injury- A Phase I Clinical Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Collaborators: Armed Forces Institute of Regenerative Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFBMTC-SCI-2013
Record Dates: First submitted 2015-06-18; First posted 2015-06-26 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; mesenchymal stem cells; transplantation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous mesenchymal stem cells (Experimental): use of mesenchymal stem cells as therapeutic intervention for spinal cord injury patients by autologous transplantation
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — autologous transplantation of mesenchymal stem cells in spinal cord injury patients
  Other Names: MSC

SUMMARY:
The conventional treatment of spinal cord injury (SCI) includes physical therapy and rehabilitation and in some cases may require surgical intervention. Although improved emergency care and aggressive treatment can help in preventing further damage and even restore minimal sensory functions, still a large proportion of patients suffer with prolonged disabilities. It led neurologists to search out for new treatment options for this otherwise debilitating disorder. Recent advances in research have developed a better understanding of stem cell biology especially their role in tissue repair and regeneration. Encouraging results in pre-clinical phase and limited human trials have proved that stem cells can be safely and effectively delivered to the injured site for regeneration of damaged tissue. Although a variety of cell types have been tried for their role in repair of spinal cord injury, majority of clinical trials employed stem cells taken from bone marrow especially mesenchymal stromal cells (MSC). Bone marrow MSCs are a good choice for regenerative therapies owing to advantages like ease of collection and ex-vivo culturing, immune tolerance and their ability to differentiate into a variety of cell types including neuronal lineage cells. Intravenous application or direct injection of MSCs into cerebrospinal fluid (CSF) via lumber puncture in animal models of SCI and brain trauma had shown that MSCs can migrate towards and integrate into injured spinal tissue and reduce cyst size and increase functional recovery. The literature indicates that acute, sub-acute and chronic injury can be a therapeutic target for MSC grafting. The mechanism of action may however vary among these conditions. In acute phase, MSC administration play anti-inflammatory role, while in sub-acute/chronic setting it may be used as neurostimulator and for cell bridging effect and possibly glial or neuronal cell replacement. The investigators propose a non-randomized, single group, open label, phase-I, interventional study to evaluate the safety and efficacy of intrathecal delivery of patient's own (autologous) bone marrow mesenchymal stem cells for treatment of spinal cord injury. This will include determination of functional recovery (neuro-muscular control and sensation) in the affected area and overall improvement in quality of life of the patients and also take into account any side effects, if observed.

DETAILED DESCRIPTION:
The role of regenerative therapies has gained more importance due to increased number of SCI in the wake of recent anti-terrorism operations by the armed forces and non-availability of any curative treatment for this category of patients. The promising results of preliminary clinical trials have proved that adult stem cells especially multipotent mesenchymal stromal cells can be safely injected and well tolerated and have shown functional improvement in SCI patients. The successful treatment in these patients will not only improve functional status of these otherwise debilitating patients, but can also reduce the burden on health care facilities. Mesenchymal stem cells have been shown to promote anatomical and functional recovery in animal models of SCI by promoting tissue sparing, axonal regeneration, and remyelination. Therapeutic effects of MSCs are primarily due to the secretion of soluble factors and the provision of extracellular matrix that provide protection and support repair. MSC are attractive candidates for transplantation into human patients because they can be easily harvested, expanded and banked, or derived directly from the patient allowing for autologous transplantation, obviating the need for immune suppression. In this study patients suffering from sub-acute and chronic phase of spinal cord injury shall be included. Patients will undergo detailed screening through MRI and motor and sensory assessment by ASIA score. Further evaluation will include electromyography (EMG) and tests for electroneurophysiological assessment like nerve conduction velocity (NCV) will also be done. Bone marrow aspiration will be done from iliac crest of the patients, followed by mononuclear cells (MNCs) separation by density gradient centrifugation. MNCs will be washed and cultured in tissue culture flasks. After 48 hours non-adherent cells will be removed from culture. Medium will be changed twice weekly till MSCs reach 70-80 % confluence. At that point MSCs will be harvested and after microbiological and other quality control testing the cellular preparation will be diluted to final concentration and infused by intrathecal injection.

Primary outcome measure is safety which will be determined by clinical evaluation by two independent neurologists during one month of hospital stay after receiving treatment course.

Secondary outcome measures will include American Spinal Injury Association (ASIA) impairment scale and NCV/EMG.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from sub-acute and chronic phase of spinal cord injury
* Traumatic spinal cord injury at the thoracic level
* American Spinal Injury Association (ASIA) impairment scale "A"
* Confirmation by MRI of injury level
* Time between injury and enrollment greater than 2 weeks
* Ability to provide informed consent

Exclusion Criteria:

* Axonic brain injury
* Inability to provide consent
* Open injuries
* Active infectious diseases
* Terminal patients
* Neurodegenerative diseases
* Evidence of meningitis
* Cerebral palsy
* Primary haematologic diseases
* Coagulopathies
* Pregnancy
* Other medical complications that contra-indicate surgery, including major respiratory complications
* Use of metal implants close to vascular structures (such as cardiac pacemaker or prosthesis) that contraindicate MRI.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 1 month
  Number of adverse events occurring in given time frame shall be reported to evaluate overall safety of the procedure

SECONDARY OUTCOMES:
Sensory and motor strength | 1 year
  Improvement in sensitivity and motor strength will be measured through change in American Spinal Injury Association (ASIA) score from baseline
Functional Independence | 1 year
  Functional Independence will be measured by FIM scoring
Muscle strength assessment | 1 year
  Shall be done using Frankel scale

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Ahmed, Principal Investigator — Commandant Armed Forces Bone Marrow Transplant Center
Locations (1):
- Armed Forces Bone Marrow Transplant Centre, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Legos JJ, Gopez JJ, Young WF. Non-surgical management of spinal cord injury. Expert Opin Investig Drugs. 2002 Apr;11(4):469-82. doi: 10.1517/13543784.11.4.469. PMID 11922856
- [Background] Zhang HT, Cheng HY, Cai YQ, Ma X, Liu WP, Yan ZJ, Jiang XD, Xu RX. Comparison of adult neurospheres derived from different origins for treatment of rat spinal cord injury. Neurosci Lett. 2009 Jul 24;458(3):116-21. doi: 10.1016/j.neulet.2009.04.045. Epub 2009 Apr 24. PMID 19394407
- [Background] Mackay-Sim A, St John JA. Olfactory ensheathing cells from the nose: clinical application in human spinal cord injuries. Exp Neurol. 2011 May;229(1):174-80. doi: 10.1016/j.expneurol.2010.08.025. Epub 2010 Sep 9. PMID 20832402
- [Background] Hernandez J, Torres-Espin A, Navarro X. Adult stem cell transplants for spinal cord injury repair: current state in preclinical research. Curr Stem Cell Res Ther. 2011 Sep;6(3):273-87. doi: 10.2174/157488811796575323. PMID 21476980
- [Background] Tetzlaff W, Okon EB, Karimi-Abdolrezaee S, Hill CE, Sparling JS, Plemel JR, Plunet WT, Tsai EC, Baptiste D, Smithson LJ, Kawaja MD, Fehlings MG, Kwon BK. A systematic review of cellular transplantation therapies for spinal cord injury. J Neurotrauma. 2011 Aug;28(8):1611-82. doi: 10.1089/neu.2009.1177. Epub 2010 Apr 20. PMID 20146557
- [Background] Karamouzian S, Nematollahi-Mahani SN, Nakhaee N, Eskandary H. Clinical safety and primary efficacy of bone marrow mesenchymal cell transplantation in subacute spinal cord injured patients. Clin Neurol Neurosurg. 2012 Sep;114(7):935-9. doi: 10.1016/j.clineuro.2012.02.003. Epub 2012 Mar 30. PMID 22464434
- [Background] Dasari VR, Veeravalli KK, Dinh DH. Mesenchymal stem cells in the treatment of spinal cord injuries: A review. World J Stem Cells. 2014 Apr 26;6(2):120-33. doi: 10.4252/wjsc.v6.i2.120. PMID 24772239
- [Background] All AH, Gharibani P, Gupta S, Bazley FA, Pashai N, Chou BK, Shah S, Resar LM, Cheng L, Gearhart JD, Kerr CL. Early intervention for spinal cord injury with human induced pluripotent stem cells oligodendrocyte progenitors. PLoS One. 2015 Jan 30;10(1):e0116933. doi: 10.1371/journal.pone.0116933. eCollection 2015. PMID 25635918
- [Derived] Satti HS, Waheed A, Ahmed P, Ahmed K, Akram Z, Aziz T, Satti TM, Shahbaz N, Khan MA, Malik SA. Autologous mesenchymal stromal cell transplantation for spinal cord injury: A Phase I pilot study. Cytotherapy. 2016 Apr;18(4):518-22. doi: 10.1016/j.jcyt.2016.01.004. PMID 26971680